CLINICAL TRIAL: NCT04176315
Title: Usability and Effectiveness of ReHub in Patients After Total Hip Arthroplasty
Acronym: REHIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Bio-Sensing Solutions S.L. (DyCare) (Industry)
Collaborators: University of Turin, Italy (Other); Presidio Sanitario San Camillo, Turin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCEB07072019
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Rehabilitation Group (Active Comparator): Participants follow the usual exercise plan designed at Presidio San Camillo for Total Hip Arthroplasty autonomously
  Interventions: Other: Conventional Home-based Rehabilitation Plan
- ReHub Group (Experimental): Participants follow the usual exercise plan designed at Presidio San Camillo for Total Hip Arthroplasty but use the telerehabilitation platform ReHub to do the exercises at home and to have their progress monitored.
  Interventions: Device: ReHub Home-based Rehabilitation Plan

INTERVENTIONS:
Other: Conventional Home-based Rehabilitation Plan — Usual intervention at Presidio Sanitario San Camillo for post-operative rehabilitation of THA patients. Participants receive inpatient care and rehabilitation for 2 weeks. At discharge, they receive a 5-exercise home-based rehabilitation plan. For the sake of homogeneity of all participants, they receive from 2 to 4 of training prior to discharge. At home, participants shall perform the exercises in the rehabilitation plan daily.
  Arms: Conventional Rehabilitation Group
Device: ReHub Home-based Rehabilitation Plan — Combination of the usual intervention at Presidio Sanitario San Camillo for post-operative rehabilitation of THA patients with ReHub, a telerehabilitation platform that serves as a guide to perform the TKA rehabilitation exercises.
  Participants receive inpatient care and rehabilitation at San Camillo for 2 weeks. At discharge, a 5-exercise home-based rehabilitation plan is carried out by a site physiotherapist by using ReHub to acquire the participant's movement pattern with a wearable inertial sensor. Participants receive from 2 to 4 sessions of ReHub prior to discharge.
  At home, participants shall perform the exercises in the rehabilitation plan with ReHub daily. The wearable inertial sensor participants must wear tracks movement while they do the TKA rehabilitation exercises. Movement is analysed and feedback is given in real time. Participants can select if they have felt pain in a scale from 1 to 10. A physiotherapist monitors the participants' progress remotely.
  Arms: ReHub Group

SUMMARY:
This is a randomized, non-blinded, parallel assignment, clinical trial for the evaluation of usability and effectiveness of ReHub, a telerehabilitation system made up of a cloud platform and an exercise kit with smart sensors, for performing rehabilitation exercises after a primary Total Hip Arthroplasty (THA).

Patients admitted to Presidio San Camillo after a THA surgery are randomly allocated to the control arm or the experimental arm with a 1:1 ratio. Participants in both arms receive inpatient care and rehabilitation for 2 weeks at San Camillo. At discharge, they are prescribed with the same daily plan of 5 exercises for autonomous home-based rehabilitation. The experimental arm participants use ReHub to do their exercises instead of working independently and physiotherapists monitor their performance and adherence remotely.

Outcomes assessment is performed at San Camillo admission (baseline), at San Camillo discharge (2 weeks from baseline) and 3 weeks after San Camillo discharge (5 weeks from baseline).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and accept the clinical study procedure and to sign an informed consent form
* Good familiarity with the Italian language
* Good predisposition to the use of technology or availability of a caregiver providing technological support to the patient
* Availability to move to the Rehabilitation Center for control visits

Exclusion Criteria:

* Age <60 or >80 years
* Admission after THA revision surgery
* Contralateral hip osteoarthritis severely limiting patient mobility and ability to comply with a rehabilitation program
* Aphasia, dementia, or psychiatric comorbidity interfering with communication or adherence to the rehabilitation process
* Respiratory, cardiac, metabolic, or other condition limiting patient mobility and ability to comply with a rehabilitation program
* Major medical complications occurring after surgery that prevented the discharge of the patient within 10 days after the surgery
* Body mass index >35kg/m2

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Change in the Timed Up-and-Go test score (s) | Baseline, 2 weeks and 5 weeks from baseline
  The TUG test outcome is the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down as the score.

SECONDARY OUTCOMES:
Change in Hip Flexion Range of Motion (º) | Baseline, 2 weeks and 5 weeks from baseline
  Range of motion of the replaced hip for flexion, without the aid of the outcomes assessor, is measured with a conventional goniometer.
Change in Hip Extension Range of Motion (º) | Baseline, 2 weeks and 5 weeks from baseline
  Range of motion of the replaced hip for extension, without the aid of the outcomes assessor, is measured with a conventional goniometer.
Change in Hip Abduction Range of Motion (º) | Baseline, 2 weeks and 5 weeks from baseline
  Range of motion of the replaced hip for abduction, without the aid of the outcomes assessor, is measured with a conventional goniometer.
Change in Quadriceps Strength (kg) | Baseline, 2 weeks and 5 weeks from baseline
  Strength of the quadriceps in the intervened leg is measured with a dynamometer.
Change in Extension Strength (kg) | Baseline, 2 weeks and 5 weeks from baseline
  Strength of the intervened leg while performing an extension movement is measured with a dynamometer.
Change in Abduction Strength (kg) | Baseline, 2 weeks and 5 weeks from baseline
  Strength of the intervened leg while performing an abduction movement is measured with a dynamometer.
Change in Self-Reported Pain Level at Rest: Numerical Rating Scale | Baseline, 2 weeks and 5 weeks from baseline
  The pain level of the intervened hip at rest is reported by the participant with a Numerical Rating Scale from 0 to 10, with 0 being the absence of pain and 100 being the worst possible pain.
Change in Self-Reported Pain Level in Movement: Numerical Rating Scale | Baseline, 2 weeks and 5 weeks from baseline
  The pain level of the intervened hip in movement is reported by the participant with a Numerical Rating Scale from 0 to 10, with 0 being the absence of pain and 100 being the worst possible pain.
Change in Hip disability and Osteoarthritis Outcome Score (HOOS) | Baseline, 2 weeks and 5 weeks from baseline
  Scores for the HOOS questionnaire range from 0% to 100%, with 0 being the worst possible score and 100 the best possible score.
Change in Functional Independence Measure (FIM) score | Baseline, 2 weeks and 5 weeks from baseline
  Scores for the FIM questionnaire range from 18 to 126, with 13 being the worst possible score and 100 the best possible score. Individual items (18) are scored from 1 (worst) to 7 (best).
Global Rating Of Change | 5 weeks from baseline
  The participant will report their perception of change from the start to the end of the study with a number from 1 (substantial worsening) to 6 (total recovery).
Satisfaction with ReHub: System Usability Scale | 5 weeks from baseline
  Measured with the score from the System Usability Scale questionnaire, which can range from 0 (worst result) to 100 (best result). Only for participants in the experimental arm.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Alessandro Minetto, Principal Investigator — University of Turin, Department of Surgical Sciences
Locations (1):
- Presidio Sanitario San Camillo, Turin, Piedmont, Italy

REFERENCES:
- [Derived] Busso C, Castorina G, Di Monaco M, Rodriguez D, Mahdavi H, Balocco S, Trucco M, Conti M, Castagna A, Minetto MA. Effectiveness of a home-based telerehabilitation system in patients after total hip arthroplasty: study protocol of a randomized controlled trial. Trials. 2020 Oct 14;21(1):852. doi: 10.1186/s13063-020-04791-4. PMID 33054811